CLINICAL TRIAL: NCT03658382
Title: Randomized Controlled Trial Evaluating Patient Satisfaction With Virtual Visits for Results Disclosure in the Brigham and Women's Hospital Cardiovascular Genetics Program
Brief Title: Virtual Visits for Results Disclosure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Noreen Kelly, Cardiovascular Medicine Fellow, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017P000434
Record Dates: First submitted 2018-09-01; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Results Disclosure (No Intervention)
- Virtual Visit Results Disclosure (Experimental)
  Interventions: Other: Virtual Visit

INTERVENTIONS:
Other: Virtual Visit — Patients will receive the results of their genetic testing via a virtual visit.
  Arms: Virtual Visit Results Disclosure

SUMMARY:
As part of this study patients who have undergone genetic testing in the Brigham and Women's Hospital Cardiovascular Genetics program will be randomized to receive the results of their genetic testing either by telephone call or virtual visit. At the completion of the telephone call or virtual visit patients will receive a survey to assess their understanding of their results and their satisfaction with their care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing genetic testing at BWH Cardiovascular Genetics clinic

Exclusion Criteria:

* Reside outside of Massachusetts
* Telephone or internet access unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | within 7 days of results disclosure
  Web-based survey focused on patient comprehension and satisfaction

IPD SHARING:
Plan to Share IPD: No
No plan to share data